CLINICAL TRIAL: NCT03595774
Title: Dose-response Effect of Dietary Nitrate on Muscle Function in Older Individuals
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Andrew Coggan, Associate Professor, Indiana University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 1712606816
Record Dates: First submitted 2018-07-11; First posted 2018-07-23 (Actual); Results first posted 2024-07-29 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-02

CONDITIONS: Aging; Sarcopenia
Keywords: nitric oxide
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Intervention Model Description: Double-blind, placebo-controlled, crossover
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Placebo (Placebo Comparator): 3.3 mL/kg concentrated beet root juice *depleted of nitrate* Other names: Beet It Sport Nitrate 400 placebo
  Interventions: Dietary Supplement: Beet root juice
- low nitrate (Active Comparator): 1.55 mL/kg concentrated beet root juice depleted of nitrate + 1.55 mL/kg concentrated beet root juice *depleted of nitrate*
  Other names: Beet It Sport Nitrate 400 placebo + Beet It Sport Nitrate 400
  Interventions: Dietary Supplement: Beet root juice
- high nitrate (Active Comparator): 3.3 mL/kg concentrated beet root juice containing nitrate
  Other names:Beet It Sport Nitrate 400
  Interventions: Dietary Supplement: Beet root juice

INTERVENTIONS:
Dietary Supplement: Beet root juice — Beet root juice
  Other Names: Beet It Sport Nitrate 400

SUMMARY:
Nitrate is a naturally-occurring substance found in foods, especially green leafy vegetables and beets. Increasing nitrate intake (by drinking beetroot juice (BRJ) has been shown to improve muscle function young and middle-aged subjects, athletes, and patients with heart failure. The purpose of this study is to determine whether dietary nitrate provides a similar benefit in older individuals, and if so, the optimal dose. We will be comparing the effects of ingesting BRJ containing a smaller or greater amount of nitrate versus the effects of a placebo (BRJ from which the nitrate has been removed).

DETAILED DESCRIPTION:
This study consists of four visits that will take a minimum of 15 days to complete.

Study Visit One (Screening) 1-2 hours The purpose of the screening visit is to explain all aspects of the study. The investigators will also determine if individuals can participate in the study. Eligible subjects will undergo a complete medical history and physical exam. They will have their blood drawn, and will provide a urine sample (to determine if they are pregnant). Subjects will also practice the entire neuromuscular function exercise test. During this test, the strength of the subject's muscles will be determined by having them kick, push and/or pull back as hard as they can while their leg is strapped to an exercise device. Blood pressure and heart rate and rhythm will be monitored.

Subjects will be instructed to consume their normal diet throughout the study. However, they will be asked to avoid eating foods high in nitrate such as beets, spinach, and collard greens the evening before each visit. They will be asked to refrain from the use of antibacterial mouthwash, such as Listerine or Cepacol, during the study. Subjects will also be asked to not chew gum or to consume alcohol or food and drinks that contain caffeine for 24 hour before each visit. This includes coffee, tea, chocolate and soft drinks such as Mountain Dew. Finally, they will be asked to fast for 12 hour prior to each study visit.

Study Visit Two - Approximately 5 hours At the beginning of this visit a catheter (small, flexible, sterile plastic tube) will be placed through a vein in one of the subject's arms. This is for collection of blood samples. Blood will be drawn four times during this visit. Each draw will be 6mL or about 1.2 teaspoons. The first blood draw will check nitrate and nitrogen levels. Subjects will then have a breath test to check nitric oxide. They will then drink about 280 mL (about 1 cup) of BRJ. In one trial, this will be a placebo, that is, BRJ from which the essentially all of the nitrate has been removed. In another trial, they will drink BRJ still containing nitrate. In a third trial, they will drink an equal mixture of the placebo and nitrate-containing BRJ. Blood and breath samples will be obtained every hour. Heart rate and blood pressure will be measured at the same times the blood and breath samples are obtained. About 2 hours after ingestion of BRJ (or placebo) subjects will be asked to perform the neuromuscular function test that was practiced during the screening visit. After completing the exercise test one final blood and breath sample will be obtained.

Study Visits Three and Four

The same procedures completed during Study Visit Two will be performed. The order of treatment (placebo vs. lower dose vs. higher dose of nitrate) will be randomized using a computer program. Neither the subjects nor the investigators will know the treatment they receive during each visit until the entire study is completed.

ELIGIBILITY:
Inclusion Criteria:

• In good health, as determined by the investigator's review of history (provided by subject at screening visit), physical examination, and routine blood and urine tests (done at screening visit)

Exclusion Criteria:

* Men and women <65 or >79 years of age
* Unable to provide informed consent
* Currently pregnant or lactating (given the age range for the study, verbal confirmation by subject is believed to be sufficient)
* Current smokers
* Significant orthopedic limitations or other contraindications to strenuous exercise
* Those taking phosphodiesterase inhibitors (e.g., Viagra)
* Those taking proton pump inhibitors, antacids, xanthine oxidase inhibitors, or on hormone replacement therapy
* Those taking anti-coagulants (e.g., Coumadin) or on anti-platelet therapy
* History of neuromuscular disease (e.g., cervical spondylotic radiculomyelpathy, lumbar spondylosis, amyotrophic lateral sclerosis, Guillain-Barré syndrome, and acquired demyelinating polyneuropathies), cardiovascular disease (e.g., > stage I hypertension, heart failure, myocardial infarction/ischemia, significant myocardial or pericardial diseases (e.g. amyloidosis, constriction), moderate or severe valvular disease, renal disease, liver disease, or anemia

Ages: 65 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 13 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew R Coggan, PhD, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Indiana University School of Health and Human Sciences, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Coggan AR. Dietary Nitrate and Muscle Function in Humans: Acute versus Chronic Mechanisms. Med Sci Sports Exerc. 2018 Apr;50(4):874. doi: 10.1249/MSS.0000000000001489. No abstract available. PMID 29547495
- [Background] Coggan AR, Broadstreet SR, Mahmood K, Mikhalkova D, Madigan M, Bole I, Park S, Leibowitz JL, Kadkhodayan A, Thomas DP, Thies D, Peterson LR. Dietary Nitrate Increases VO2peak and Performance but Does Not Alter Ventilation or Efficiency in Patients With Heart Failure With Reduced Ejection Fraction. J Card Fail. 2018 Feb;24(2):65-73. doi: 10.1016/j.cardfail.2017.09.004. Epub 2017 Sep 12. PMID 28916479
- [Background] Coggan AR, Peterson LR. Dietary Nitrate and Skeletal Muscle Contractile Function in Heart Failure. Curr Heart Fail Rep. 2016 Aug;13(4):158-65. doi: 10.1007/s11897-016-0293-9. PMID 27271563
- [Background] Rimer EG, Peterson LR, Coggan AR, Martin JC. Increase in Maximal Cycling Power With Acute Dietary Nitrate Supplementation. Int J Sports Physiol Perform. 2016 Sep;11(6):715-720. doi: 10.1123/ijspp.2015-0533. Epub 2016 Aug 24. PMID 26641379
- [Background] Coggan AR, Leibowitz JL, Spearie CA, Kadkhodayan A, Thomas DP, Ramamurthy S, Mahmood K, Park S, Waller S, Farmer M, Peterson LR. Acute Dietary Nitrate Intake Improves Muscle Contractile Function in Patients With Heart Failure: A Double-Blind, Placebo-Controlled, Randomized Trial. Circ Heart Fail. 2015 Sep;8(5):914-20. doi: 10.1161/CIRCHEARTFAILURE.115.002141. Epub 2015 Jul 15. PMID 26179185
- [Background] Coggan AR, Leibowitz JL, Kadkhodayan A, Thomas DP, Ramamurthy S, Spearie CA, Waller S, Farmer M, Peterson LR. Effect of acute dietary nitrate intake on maximal knee extensor speed and power in healthy men and women. Nitric Oxide. 2015 Aug 1;48:16-21. doi: 10.1016/j.niox.2014.08.014. Epub 2014 Sep 6. PMID 25199856

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Then Low Then High: 3.3 mL/kg concentrated beet root juice *depleted of nitrate* (1 day), washout (7 days), 1.55 mL/kg concentrated beet root juice containing nitrate + 1.55 mL/kg concentrated beet root juice *depleted of nitrate* (1 day), washout (7 days), 3.3 mL/kg concentrated beet root juice containing nitrate (1 day)
- Low Then High Then Placebo: 1.55 mL/kg concentrated beet root juice containing nitrate + 1.55 mL/kg concentrated beet root juice *depleted of nitrate* (1 day), washout (7 days), 3.3 mL/kg concentrated beet root juice containing nitrate (1 day), washout (7 days), 3.3 mL/kg concentrated beet root juice *depleted of nitrate* (1 day)
- High Then Placebo Then Low: 3.3 mL/kg concentrated beet root juice containing nitrate (1 day), washout (7 days), 3.3 mL/kg concentrated beet root juice *depleted of nitrate* (1 day)washout (7 days),1.55 mL/kg concentrated beet root juice containing nitrate + 1.55 mL/kg concentrated beet root juice *depleted of nitrate* (1 day)
- High Then Low Then Placebo: 3.3 mL/kg concentrated beet root juice containing nitrate (1 day), washout (7 days), 1.55 mL/kg concentrated beet root juice containing nitrate + 1.55 mL/kg concentrated beet root juice *depleted of nitrate* (1 day), washout (7 days),3.3 mL/kg concentrated beet root juice *depleted of nitrate* (1 day)
Period: Overall Study
Arm/Group | Placebo Then Low Then High | Low Then High Then Placebo | High Then Placebo Then Low | High Then Low Then Placebo
Started | 3 | 4 | 3 | 3
Completed | 2 | 3 | 2 | 2
Not Completed | 1 | 1 | 1 | 1
Not completed — Adverse Event | 1 | 0 | 1 | 0
Not completed — screen failure | 0 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- High Then Placebo Then Low: 3.3 mL/kg concentrated beet root juice containing nitrate (1 day), washout (7 days), 3.3 mL/kg concentrated beet root juice *depleted of nitrate* (1 day), washout (7 days), 1.55 mL/kg concentrated beet root juice containing nitrate + 1.55 mL/kg concentrated beet root juice *depleted of nitrate* (1 day)
- High Then Low Then Placebo: 3.3 mL/kg concentrated beet root juice containing nitrate (1 day)washout (7 days), 1.55 mL/kg concentrated beet root juice containing nitrate + 1.55 mL/kg concentrated beet root juice *depleted of nitrate* (1 day), washout (7 days), 3.3 mL/kg concentrated beet root juice *depleted of nitrate* (1 day)
- Total: Total of all reporting groups
Arm/Group | Placebo Then Low Then High | Low Then High Then Placebo | High Then Placebo Then Low | High Then Low Then Placebo | Total
Number analyzed (Participants) | 2 | 3 | 2 | 2 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 69 (4) | 72 (1) | 70 (4) | 70 (4) | 70 (3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 2 | 2 | 8
  Male | 1 | 0 | 0 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 3 | 2 | 2 | 9
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 2 | 3 | 2 | 2 | 9
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 3 | 2 | 2 | 9

OUTCOME MEASURES:

1. Primary Outcome: Maximal Knee Extensor Velocity
Description: Maximal knee extensor velocity determined using isokinetic dynamometry
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: rad/s
Groups:
- Placebo; Low Nitrate: 1.55 mL/kg concentrated beet root juice containing nitrate + 1.55 mL/kg concentrated beet root juice *depleted of nitrate* (1 day)
  Other names: Beet It Sport Nitrate 400
  Beet root juice: Beet root juice
- High Nitrate: 3.3 mL/kg concentrated beet root juice containing nitrate (1 day)
  Other names: Beet It Sport Nitrate 400
  Beet root juice: Beet root juice
Arm/Group | Placebo | Low Nitrate | High Nitrate
Number analyzed (Participants) | 9 | 9 | 9
rad/s | 10.83 (2.41) | 11.91 (2.01) | 11.24 (2.32)
Statistical Analysis 1: Comparison: Placebo vs Low Nitrate vs High Nitrate; Test type: Superiority; p = 0.0833, ANOVA — a priori threshold for statistical significance of P<0.05; One-way ANOVA for repeated measures followed by Holm-Šídák's multiple comparisons test

2. Primary Outcome: Maximal Knee Extensor Power
Description: Maximal knee extensor power determined using isokinetic dynamometry
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: W/kg
Arm/Group | Placebo | Low Nitrate | High Nitrate
Number analyzed (Participants) | 9 | 9 | 9
W/kg | 3.74 (1.19) | 3.92 (1.10) | 3.69 (1.04)
Statistical Analysis 1: Comparison: Placebo vs Low Nitrate vs High Nitrate; Test type: Superiority; p = 0.0131, ANOVA — a priori threshold for statistical significance of P<0.05; One-way ANOVA for repeated measures followed by Holm-Šídák's multiple comparisons test

3. Secondary Outcome: Plasma Nitrite
Time Frame: 0, 1, 2, 3 h after ingestion
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Placebo | Low Nitrate | High Nitrate
Number analyzed (Participants) | 9 | 9 | 9
umol/L
  0 h | .306 (.138) | 40 (16) | .341 (.165)
  1 h | .299 (.067) | .459 (.203) | .478 (.219)
  2 h | .326 (.113) | .528 (.219) | .949 (.535)
  3 h | .347 (.140) | .820 (.543) | 1.216 (.458)
Statistical Analysis 1: Comparison: Placebo vs Low Nitrate vs High Nitrate; Test type: Superiority; p = 0.012728, ANOVA — a prior threshold for significant of P<0.05; Two-way ANOVA for repeated measured followed by Holm-Šídák's multiple comparisons test

4. Secondary Outcome: Plasma Nitrate
Time Frame: 0, 1, 2, 3 h after ingestion
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Placebo | Low Nitrate | High Nitrate
Number analyzed (Participants) | 9 | 9 | 9
umol/L
  0 h | 55 (31) | 40 (16) | 34 (14)
  1 h | 57 (14) | 523 (155) | 793 (218)
  2 h | 67 (17) | 624 (158) | 1184 (266)
  3 h | 66 (16) | 628 (142) | 1296 (282)
Statistical Analysis 1: Comparison: Placebo vs Low Nitrate vs High Nitrate; Test type: Superiority; p = 0.00000002, ANOVA — a priori threshold for statistical significance of P<0.05; Two-way ANOVA for repeated measures followed by Holm-Šídák's multiple comparisons test

5. Secondary Outcome: Breath Nitric Oxide
Time Frame: 0, 1, 2, 3 h after ingestion
Measure: Mean (Standard Deviation); unit: ppm
Groups:
- Placebo: 3.3 mL/kg concentrated beet root juice *depleted of nitrate* (1 day)
  Other names: Beet It Sport Nitrate 400
  Beet root juice: Beet root juice
Arm/Group | Placebo | Low Nitrate | High Nitrate
Number analyzed (Participants) | 9 | 9 | 9
ppm
  0 h | 19 (10) | 18 (9) | 18 (8)
  1 h | 22 (10) | 39 (18) | 31 (12)
  2 h | 25 (10) | 43 (21) | 36 (12)
  3 h | 21 (11) | 50 (31) | 36 (17)
Statistical Analysis 1: Comparison: Placebo vs Low Nitrate vs High Nitrate; Test type: Superiority; p = 0.017215, ANOVA — a priori threshold for statistical significance of P<0.05; Two-way ANOVA for repeated measures followed by Holm-Šídák's multiple comparisons test

ADVERSE EVENTS:
Time Frame: 2 wk (during study participation)
Groups:
- All Study Participants/Arms: All study participants/arms
Arm/Group | All Study Participants/Arms
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-06-03): https://cdn.clinicaltrials.gov/large-docs/74/NCT03595774/Prot_SAP_000.pdf
  • Informed Consent Form (2019-12-10): https://cdn.clinicaltrials.gov/large-docs/74/NCT03595774/ICF_001.pdf